CLINICAL TRIAL: NCT01635998
Title: Adjunctive Renal Denervation to Modify Hypertension and Sympathetic Tone as Upstream Therapy in the Treatment of Atrial Fibrillation
Brief Title: Adjunctive Renal Denervation in the Treatment of Atrial Fibrillation
Acronym: H-FIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 12-1465; GCO 12-1465
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Uncontrolled Hypertension; Atrial Fibrillation
Keywords: renal sympathetic denervation; renal catheter ablation; hypertension
MeSH Terms: conditions — Atrial Fibrillation; Hypertension | interventions — Denervation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental): These subjects will undergo routine catheter ablation of atrial fibrillation PLUS renal sympathetic denervation with the Boston Scientific Vessix Renal Denervation System.
  Interventions: Device: Boston Scientific Vessix Renal Denervation System
- Control arm (No Intervention): These subjects will undergo routine catheter ablation of atrial fibrillation only.

INTERVENTIONS:
Device: Boston Scientific Vessix Renal Denervation System — Renal sympathetic denervation is modulation of the nerves which run along the renal arteries (the renal sympathetic nerves) with radiofrequency energy. This is the same energy source used to perform your heart ablation.
  Boston Scientific Vessix Renal Denervation System, Boston Scientific, Inc., Quincy, Massachusetts
  Other Names: renal denervation; denervation
  Arms: Intervention arm

SUMMARY:
The objective of the H-FIB trial is to determine the role of renal sympathetic denervation in the prevention of Atrial Fibrillation (AF) recurrence in patients with hypertension for whom a catheter-based AF ablation procedure is planned. Patients will be randomized to either AF catheter ablation (usual therapy) or AF catheter ablation plus renal sympathetic denervation.

DETAILED DESCRIPTION:
The purpose of this study is to examine the potential additional benefit of performing renal sympathetic denervation at the same time as an AF ablation procedure, in order to improve the long-term success of the AF procedure.

To take part in this study, you must meet all study requirements. Screening visit tests and procedures such as a physical exam, blood pressure, review of medical history, blood sample, and a Transthoracic Echocardiogram (TTE) are done to see if you are eligible to be in the study.

Patients who qualify for the study and provide consent will undergo catheter ablation for AF. Very thin electrode catheters, similar to long wires, will be inserted into blood vessels in the groin. Using the ablation catheter, we will "ablate" or damage the tissue adjacent to your pulmonary veins that is not behaving normally.

Immediately following the catheter ablation, patients will undergo a renal angiogram in order to assess suitability for catheter-based renal sympathetic denervation. A renal angiogram is an x-ray study of the blood vessels in the kidney to evaluate for blockage, and abnormalities that could be affecting the blood supply to the kidney. It is performed by injecting contrast dye through a catheter (a tiny tube) into the blood vessels of the kidney.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria
* Age ≥ 18 years of age
* History of AF (paroxysmal or persistent) and planned for a guideline-supported catheter ablation procedure
* History of significant hypertension (defined as SBP ≥160 mm Hg and/or DBP ≥100 mmHg) and receiving treatment with at least one anti-hypertensive medication OR Clinical History of hypertension and receiving treatment with at least two anti-hypertensive medications (specifically for blood pressure reduction).
* Renal vasculature is accessible as determined by intra-procedural renal angiography.
* Ability to understand the requirements of the study
* Willingness to adhere to study restrictions, comply with all post-procedural follow-up requirements and to sign informed consent

Exclusion Criteria

* Inability to undergo AF catheter ablation (e.g., presence of a left atrial thrombus, contraindication to all anticoagulation)
* Prior left atrial ablation for an atrial arrhythmia (before this index procedure)
* Patients with NYHA class IV congestive heart failure
* Individual has known secondary hypertension
* Individual has renal artery anatomy that is ineligible for treatment including:

  1. Inability to access renal vasculature
  2. Main renal arteries < 3 mm in diameter or < 20 mm in length.
  3. Hemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery which, in the eyes of the operator, would interfere with safe cannulation of the renal artery or meets standards for surgical repair or interventional dilation.
  4. A history of prior renal artery intervention including balloon angioplasty or stenting that precludes a possibility of ablation treatment.
* Individual has an estimated glomerular filtration rate (eGFR) of less than 45mL/min/1.73m2, using the MDRD calculation.
* Individual has a single functioning kidney (either congenitally or iatrogenically).
* Individual is pregnant or nursing.
* Life expectancy <1 year for any medical condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (8):
- United States (6):
  - Regional Cardiology Associates, Sacramento, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
- Na Homolce Hospital, Prague, Czechia
- Siberian Biomedical Research Center Ministry of Health Russian Federation, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Renal Sympathetic Denervation PLUS Catheter Ablation: Routine catheter ablation of atrial fibrillation PLUS renal sympathetic denervation with the Boston Scientific Vessix Renal Denervation System.
  Boston Scientific Vessix Renal Denervation System: Renal sympathetic denervation is modulation of the nerves which run along the renal arteries (the renal sympathetic nerves) with radiofrequency energy. This is the same energy source used to perform your heart ablation.
- Routine Catheter Abation: Routine catheter ablation of atrial fibrillation only.
Period: Overall Study
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Started | 28 | 22
Completed | 24 | 15
Not Completed | 4 | 7
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (6.9) | 65.3 (8.2) | 65.17 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 22 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 22 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Type of Atrial Fibrillation (AF) [Count of Participants; unit: Participants]
  Paroxysmal AF | 20 | 15 | 35
  Persistent AF | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Anti-arrhythmic Drug (AAD)-Free Single-procedure Freedom From Atrial Fibrillation Recurrence
Description: The primary endpoint of this study is anti-arrhythmic drug (AAD)-free single-procedure freedom from AF recurrence through 12 months (not including a 90 day blanking period).
Time Frame: up to 12 months
Measure: Number; unit: recurrences
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
recurrences | 6 | 2

2. Secondary Outcome: AAD-free Single-procedure Freedom From AF Recurrence
Description: AAD-free single-procedure freedom from AF recurrence through 24 months (not-including recurrences within the first 90 days of the initial ablation procedure)
Time Frame: up to 24 months
Measure: Number; unit: recurrences
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
recurrences | 7 | 6

3. Secondary Outcome: Freedom From AF Recurrence Despite Taking AADs
Description: Freedom from AF recurrence through 24 months (not-including the pre-defined 90 day blanking period) despite taking AADs
Time Frame: up to 24 months
Measure: Number; unit: recurrences
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
recurrences | 6 | 5

4. Secondary Outcome: Blood Pressure Control as Compared to Baseline
Description: Blood pressure control between the two groups as compared to baseline at 6 months, 12 months and 24 months.
Time Frame: baseline, 6 months, 12 months, and 24 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
mmHg
  Systolic Baseline | 146.6 (20.6) | 143.45 (18.47)
  Systolic 6 months | 136.88 (17.36) | 142.06 (78.94)
  Systolic 12 months | 137.88 (17.55) | 144.53 (21.6)
  Systolic 24 months | 133.88 (14.4) | 138.7 (19.9)
  Diastolic Baseline | 81.46 (13.4) | 79.18 (12.45)
  Diastolic 6 months | 80.88 (10.08) | 78.94 (7.8)
  Diastolic 12 months | 82.36 (9.19) | 82.03 (6.6)
  Diastolic 24 months | 79.8 (7.48) | 78.87 (9.75)

5. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: Number of Participants with Major adverse cardiac events (MACE) defined as a non-weighted composite score of: death, stroke, CHF hospitalization, and clinically diagnosed thromboembolic events other than stroke and hemorrhage requiring transfusion within 12 months of randomization
Time Frame: within 12 months of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
Participants | 0 | 1

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: SAE-any experience that results in a fatality or is life threatening; results in significant or persistent disability; requires or prolongs hospitalization; results in congenital anomaly/birth defect; or represents other significant hazards or potentially serious harm to research subjects or others, in the opinion of the investigators. Important medical events that may not result in above may be considered a SAE when, based upon appropriate medical judgment, they may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
Participants | 5 | 1

7. Secondary Outcome: Left Atrial (LA) Size
Description: LA size by TTE at baseline and at 12 months
Time Frame: at baseline and at 12 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
cm
  Baseline | 5.4 (0.8) | 4.7 (1.3)
  12 months | 5.19 (0.9) | 4.68 (1.4)

8. Secondary Outcome: Ejection Fraction (EF)
Description: Ejection fraction (EF) is a measurement, expressed as a percentage, of how much blood the left ventricle pumps out with each contraction. A normal heart's ejection fraction may be between 50 and 70 percent.
Time Frame: at baseline and at 12 months
Measure: Mean (Standard Deviation); unit: percent of blood
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
percent of blood
  Baseline | 62.52 (6.88) | 63.84 (6.25)
  12 months | 62.9 (7.21) | 64.5 (4.53)

9. Secondary Outcome: Number of Participants With Procedure Adverse Events
Description: Causality will be defined as adverse events that, after careful medical evaluation, are considered with a high degree of certainty to be related to the intervention (AF ablation ± renal sympathetic denervation).
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
Participants | 6 | 1

10. Secondary Outcome: Number of Anti-hypertensive Medications
Description: Total number of anti-hypertensive medications at study end, compared between the two treatment arms
Time Frame: baseline and 24 months
Measure: Mean (Standard Deviation); unit: medications
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
medications
  Baseline | 2.8 (0.95) | 2.5 (1.0)
  24 months | 2.8 (1.0) | 2.35 (1.0)

11. Secondary Outcome: Atrial Fibrillation Effect on QualiTy-of-life Questionnaire (AFEQT)
Description: The change in quality of life (QoL) from baseline to 12 months as measured by AFEQT, a 20- item instrument. Full range from 0 to 100, with higher score indicates higher level of QoL.
Time Frame: baseline, 12 months and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Renal Sympathetic Denervation PLUS Catheter Ablation | Routine Catheter Abation
Number analyzed (Participants) | 28 | 22
score on a scale
  Baseline | 72.75 (22.85) | 75.4 (26.54)
  12 months | 37.95 (16.13) | 30 (11.58)
  24 months | 39.8 (20.32) | 36.57 (21.1)

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- Catheter Ablation of Atrial Fibrillation PLUS Renal Sympatheti: Routine catheter ablation of atrial fibrillation PLUS renal sympathetic denervation with the Boston Scientific Vessix Renal Denervation System.
  Boston Scientific Vessix Renal Denervation System: Renal sympathetic denervation is modulation of the nerves which run along the renal arteries (the renal sympathetic nerves) with radiofrequency energy. This is the same energy source used to perform your heart ablation.
Arm/Group | Catheter Ablation of Atrial Fibrillation PLUS Renal Sympatheti | Routine Catheter Abation
All-Cause Mortality (participants affected / at risk) | 1/28 | 1/22
Serious Adverse Events (participants affected / at risk) | 12/28 | 4/22
Other Adverse Events (participants affected / at risk) | 6/28 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Catheter Ablation of Atrial Fibrillation PLUS Renal Sympatheti (N=28) | Routine Catheter Abation (N=22)
Bleeding (Blood and lymphatic system disorders) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac Arrhythmia (Congenital, familial and genetic disorders) | 1 | 0
Enlarged Prostate (Renal and urinary disorders) | 0 | 1
Esophageal Ulcer (Gastrointestinal disorders) | 1 | 0
Femoral Pseudoaneurysm (Vascular disorders) | 3 | 0
Fever (Immune system disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutropenic fever (Immune system disorders) | 1 | 0
Pulmonary Edema (General disorders) | 0 | 1
Renal Dysfunction (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Catheter Ablation of Atrial Fibrillation PLUS Renal Sympatheti (N=28) | Routine Catheter Abation (N=22)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Aortic Aneurysm Dissection (Cardiac disorders) | 0 | 1
Atypical Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bleeding (Blood and lymphatic system disorders) | 0 | 2
Blurred vision (Eye disorders) | 1 | 0 — Left eye
Groin Hematoma (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Skin and subcutaneous tissue disorders) | 1 | 0
Hemoptysis (Gastrointestinal disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — pain after popping from jerking motion
Syncope (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT01635998/Prot_SAP_000.pdf